CLINICAL TRIAL: NCT01396538
Title: Prevalence of Occult HBV Infection Among Anti-HBc Alone Group in Northern Taiwan
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Yi-Kuei Chen, doctor, Taipei Medical University WanFang Hospital
Other Study IDs: 100028
Record Dates: First submitted 2011-07-04; First posted 2011-07-18 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: HBV Coinfection
Keywords: anti-HBc alone ；occult HBV infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Atni-HBs to HBsAg and Anit-HBc was interpreted based on three hepatitis markers for clinical detection of HBV-infections. HBAg and Anti-HBs were negative and the Anit-HBc-positive referred to as Anti-HBc alone. When the Anti-HBc alone occurs, patients may be due to mutations in HBV HBsAg can not be detected due to (1), but if by the molecular diagnostics by polymerase chain reaction (PCR) technology can detect HBV DNA present. When Anti-HBc alone in patients with serum HBV DNA can be measured, then there may be occult HBV infection. In different countries, Occult HBV infection in the Anti-HBc Alone group had significant differences in the prevalence (2.9 ~ 22.8%) (2), but prevalence survey in Taiwan there are very few studies on this , It is hoped to be able to investigation the prevalence of occult HBV infection Among Anti-HBc Alone.

DETAILED DESCRIPTION:
The main use of this program, Taipei Medical University - Wan Fang Hospital in clinical specimens using the Roche system (Corbas e601) operating HBsAg, Anti-HBs, Anti-HBc to screen for the Anti-HBc alone group. Recycling Roche molecular system (Taq48) Real-time PCR to detect all anti-HBc alone population to understand their serum HBV-DNA viral load, in order to understand Occult HBV infection in the Anti-HBc alone group, the prevalence and viral load changes in these studies through the clinical units to provide occult HBV infection as a reference basis.

ELIGIBILITY:
Inclusion Criteria:

HBsAg(-)；Anti-HBs(-)；Anti-HBc(+)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: anti-HBc alone（HBsAg(-)；Anti-HBs(-)；Anti-HBc(+)）；occult HBV infection（the presence of HBV DNA in the liver and blood, in the absence Occult HBV of detectable HBsAg
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-06; Study Completion 2012-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Kue Chen, college, Study Director — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan, Taiwan